CLINICAL TRIAL: NCT05579353
Title: The Roles and Molecular Mechanism of Exosomal Circ-LRBA That Regulates miR-451/CRTC2 Signaling Axis in Colorectal Cancer Progression
Brief Title: The Roles of Exosomal Circ-LRBA and 451/CRTC2 Signaling Axis in Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Jingbo Chen (Other)
Responsible Party: Sponsor-Investigator, Jingbo Chen, Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2022
Record Dates: First submitted 2022-10-09; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cancer group
  Interventions: Other: nothing
- control group
  Interventions: Other: nothing

INTERVENTIONS:
Other: nothing — nothing

SUMMARY:
Colorectal cancer (CRC) is one of the most common malignant tumors in the world. Most of the patients with colorectal cancer were diagnosed in poor stage. Although 40% to 50% patients of colorectal cancer can be cured by surgery, but most patients have undergent metastasis or recurrence, and eventually death. In recent years, molecular targeted therapy has shown significant efficacy in specific patients. It was necessary to detect the corresponding molecular targets of tumors before selecting appropriate targeted drugs in clinic. The changing state of related gene molecules in colorectal cancer played a key role in drug selection, there were few effective targets so far. At present, metastasis and recurrence still be the most difficult problems in treatment. Therefore, investigators should deeply study the occurrence and development of colorectal cancer at the gene level and look for new biomarkers to predict the prognosis. Furthermore, the study can clarify the exact molecular mechanism of colorectal cancer. These will be important clinical significance for targeted therapy of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1.18-80 years old.

2.18.5 < BMI < 27.9.

3. The surgical methods are radical resection of rectal cancer, resection of right colon cancer, resection of left colon cancer and radical resection of sigmoid colon cancer.

Exclusion Criteria:

1. Those who refuse to collect samples.
2. Patients with severe dysfunction of coagulation, hepatorenal dysfunction or severe cardiopulmonary diseases.
3. Patients who has a history of neoadjuvant radiotherapy or chemotherapy.
4. Combining with distant multiple metastases of tumor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
expressional quantity | Through study completion, an average of 2 year
  Expression of CRTC2 in patient samples

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Lixia, China

IPD SHARING:
Plan to Share IPD: Yes